CLINICAL TRIAL: NCT00125112
Title: Internet Weight Control for Bingeing Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK65757 (completed)
Record Dates: First submitted 2005-07-28; First posted 2005-07-29 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Obesity; Eating Disorders
Keywords: binge eating; weight loss; obesity
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders; Bulimia; Weight Loss

INTERVENTIONS:
Behavioral: Internet-based intervention designed to reduce binge eating and improve healthy weight regulation

SUMMARY:
The purpose of this study is to determine if an internet-based intervention designed to reduce binge eating and improve healthy weight regulation skills will result in reductions in binge eating and weight loss, or weight maintenance, in overweight adolescents who binge eat.

DETAILED DESCRIPTION:
The purpose of this study is to determine if an internet-based intervention designed to reduce binge eating and improve healthy weight regulation skills will result in reductions in binge eating and weight loss, or weight maintenance, in overweight adolescents who binge eat.

ELIGIBILITY:
Inclusion Criteria:

* Female and male high school students in Hayward Unified School District or Meridian School District
* 85th or greater percentile for age-adjusted weight
* Objective binge eating one or more times weekly for a duration of ≥ 3 months
* Access to a computer with internet access
* English literacy at a sixth grade reading level

Exclusion Criteria:

* Current (or history of) diagnosis of anorexia or bulimia nervosa
* Active suicidal ideation
* Current enrollment in a formal weight loss or binge eating program (e.g., Weight Watchers)
* Any medical condition in which the actual condition or treatment affects weight and/or appetite (i.e., cancer, diabetes)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-02; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Frequency of binge eating; weight

CONTACTS AND LOCATIONS:
Overall Officials: C. Barr Taylor, M.D., Principal Investigator — Stanford University Department of Psychiatry and Behavioral Sciences
Locations (1):
- Stanford University Department of Psychiatry and Behavioral Sciences, Stanford, California, United States

REFERENCES:
- [Derived] Jones M, Luce KH, Osborne MI, Taylor K, Cunning D, Doyle AC, Wilfley DE, Taylor CB. Randomized, controlled trial of an internet-facilitated intervention for reducing binge eating and overweight in adolescents. Pediatrics. 2008 Mar;121(3):453-62. doi: 10.1542/peds.2007-1173. PMID 18310192